CLINICAL TRIAL: NCT05453006
Title: Reducing Cervical Cancer Screening Disparities in Somali Immigrant Women Through a Primary Care-based HPV Self-sampling Intervention
Brief Title: HPV Self-Sampling in Somali Women (Isbaar Project)
Acronym: Isbaar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FMCH-2019-27849
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Papillomavirus Infection; Uterine Diseases; Uterine Cervical Disease
Keywords: DNA virus infections; virus diseases; infections; tumor virus infections; papilloma; uterine diseases; uterine cervical diseases; Somali women; primary care; cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Uterine Diseases; Uterine Cervical Diseases; DNA Virus Infections; Virus Diseases; Infections; Tumor Virus Infections; Papilloma

STUDY DESIGN:
Intervention Model Description: Hybrid Type 2 effectiveness-implementation study; difference-in-difference methods to compare between-period changes in 3 intervention and Fairview non-intervention clinics.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): At the three intervention clinics, clinic providers or staff will offer women the option to perform HPV self-sampling as an alternative to cervical cancer screening by a clinician.
  Interventions: Device: COPAN 552c.80 FLOQSwab
- Control (No Intervention): Control clinics will have passive participation and their only involvement will be that data will be pulled from these clinics. Women in the control clinics will be offered usual care cervical cancer screening by a clinician. The research team will not have any contact with women in the control clinics.

INTERVENTIONS:
Device: COPAN 552c.80 FLOQSwab — The study will implement HPV self-sampling as an option for cervical cancer screening alongside usual care for Somali women, and evaluate changes pre and post implementation, compared to Fairview non-intervention clinics.
  Arms: Intervention

SUMMARY:
This study plans to assess the effect of implementing HPV self-sampling in primary care on uptake of cervical cancer screening in 30-65 year old Somali women who are due for cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a Somali woman
* between ages of 30-65
* eligible for cervical cancer screening

Exclusion Criteria:

* Ineligible for cervical cancer screening, including having a history of cervical cancer or a hysterectomy without intact cervix

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3367 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2025-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Pratt, PhD, Principal Investigator — University of Minnesota; Rachel Winer, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Pratt R, Bliss Barsness C, Lin J, Adan F, Abdi S, Mohamed S, Farah H, Trofholz A, Desai J, Fordyce K, Ghebre R, Ibrahim A, Ramer T, Szpiro A, Weiner BJ, Yohe S, Winer RL. Experience with Cervical Cancer Screening and Views on HPV Self-Sampling Among Somali American Women. J Gen Intern Med. 2025 Dec 18. doi: 10.1007/s11606-025-10080-0. Online ahead of print. PMID 41410863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinics were assigned to study arms; 3 clinics were assigned to the intervention group and 37 clinics to the control group. However, as all data analysis is done at the participant level, we are reflecting participant data in the flow here.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1948; 3 Clinics | 1419; 37 Clinics
Completed | 1948; 3 Clinics | 1419; 37 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1948 | 1419 | 3367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1948 | 1419 | 3367
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1948 | 1419 | 3367
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1904 | 1171 | 3075
  White | 1 | 1 | 2
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 38 | 241 | 279

OUTCOME MEASURES:

1. Primary Outcome: Difference-in-difference Comparison
Description: Difference-in-difference Cox proportional hazards regression to compare screening completion changes 12-months pre- /post-implementation in intervention versus control clinics, adjusting for age, screening history, and CDC social vulnerability index (SVI).
Time Frame: Up to one-year (time-to-event) to initiate screening in each of the pre and post implementation periods.
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Groups:
- Intervention & Control Arm Participants: At the three intervention clinics, clinic providers or staff will offer women the option to perform HPV self-sampling as an alternative to cervical cancer screening by a clinician.
  Women in the 3 intervention clinics will be offered HPV self-sampling as an option for cervical cancer screening alongside usual care for Somali women, and evaluate changes pre and post implementation, compared to Fairview non-intervention clinics.
  Women in the 37 control clinics will be offered usual care cervical cancer screening by a clinician. The research team will not have any contact with women in the control clinics.
Arm/Group | Intervention & Control Arm Participants
Number analyzed (Participants) | 3367
Hazard ratio | 1.8 [1.41 to 2.32]

2. Primary Outcome: Pre-implementation Period Cervical Cancer Screening Completion
Description: For the pre-implementation period (prior to intervention clinics offering the option to perform HPV self-sampling), the operational definition of screening completion is receiving Pap and/or HPV testing by a clinician.
Time Frame: Up to one-year (time-to-event) to initiate screening in the pre-implementation period.
Population: Patients in the pre-implementation period
Measure: Number; unit: Participants who completed screening
Arm/Group | Intervention | Control
Number analyzed (Participants) | 987 | 758
Participants who completed screening | 170 | 482

3. Primary Outcome: Post-implementation Period Cervical Cancer Screening Completion.
Description: For the post-implementation period, the operational definition of screening completion accounts for hybrid options that allow for either HPV self-sampling, or Pap and/or HPV testing by a clinician. We define screening completion as:
  1. receiving Pap and/or HPV testing by a clinician;
  2. self-sampling HPV-negative or HPV16/18+; or
  3. self-sampling positive for other high-risk HPV types (i.e., "HPV+ other") or unsatisfactory and returning for a follow-up Pap test to complete the screening episode. For women with "HPV+ other" or unsatisfactory test results on self-sampling, a follow-up Pap test is required; if the Pap test is not completed within 3 months, the woman will not be considered screened.
Time Frame: Up to one-year (time-to-event) to initiate screening in the post implementation period.
Population: Patients in the post-implementation period
Measure: Number; unit: Participants who completed screening
Arm/Group | Intervention | Control
Number analyzed (Participants) | 961 | 661
Participants who completed screening | 303 | 436

ADVERSE EVENTS:
Time Frame: 12 months (post-implementation period)
Description: The pre-implementation period was observational; all adverse events are assessed in the post-implementation period.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/1948 | 0/1419
Serious Adverse Events (participants affected / at risk) | 0/1948 | 0/1419
Other Adverse Events (participants affected / at risk) | 0/1948 | 0/1419

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05453006/Prot_SAP_001.pdf
  • Informed Consent Form (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05453006/ICF_000.pdf